CLINICAL TRIAL: NCT03106298
Title: Iron Deficiency and Fibroblast Growth Factor 23 Regulation in Chronic Kidney Disease and Heart Failure
Brief Title: Iron Deficiency and FGF23 Regulation in CKD and HF
Acronym: INDIGO
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Rupal Mehta, Assistant Professor of Medicine/Nephrology, Northwestern University
Other Study IDs: STU00201742
Record Dates: First submitted 2017-03-22; First posted 2017-04-10 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Diseases; Chronic Heart Failure; Iron Deficiency Anemia
Keywords: Iron Deficiency; Fibroblast Growth Factor 23; Phosphate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be processed and stored in the study freezers with a de-identified study number and collection date.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Iron Sucrose Treatment: All patients with iron deficiency anemia (those without CKD or HF, those with CKD only, those with HF only, and those with CKD/HF) will be given 5 weekly doses of 200 mg of intravenous iron sucrose.
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Iron Sucrose — All participants will be given intravenous iron sucrose (200 mg) weekly for 5 weeks. Iron sucrose is infused over 60 minutes.
  Other Names: Venofer

SUMMARY:
This study investigates the effects of intravenous (IV) iron sucrose therapy on blood levels of Fibroblast Growth Factor 23 (FGF23, a protein that regulates the amount of phosphate in the body) in iron deficiency anemia in healthy participants, participants with Congestive Heart Failure (CHF, where the heart does not pump adequate blood supply to the body), participants with Chronic Kidney Disease (CKD, where the kidney function is reduced), and participants with CKD and CHF.

DETAILED DESCRIPTION:
Iron is a key part of our red blood cells which bring oxygen to our body's tissues. Without iron, our blood cannot carry oxygen. The body normally gets iron through diet and it also re-uses iron from old red blood cells. When iron stores are low, patients get iron deficiency anemia. This can happen because patients lose more red blood cells and iron than the body can replace, the body does not do a good job at absorbing iron from the diet, or the body is able to absorb iron but patients are not getting enough iron from their diets. Many patients with chronic diseases such as CKD and CHF also have iron deficiency anemia.

Iron deficiency may also cause a hormone in the body named FGF23 to rise. FGF23 is a hormone that is made in bone and has an important role in the heart and kidney. When the kidneys are not working properly, as in CKD, or when the heart is not pumping correctly, as in CHF, FGF23 levels in the blood go up. Many patients with CKD or CHF also have low levels of iron. In these cases, FGF23 levels may rise even more. Too much FGF23 in the blood may lead to an increased risk of heart problems and accelerate loss of kidney function. The best way to control FGF23 levels in the blood in CKD and CHF is not known.

The investigators are conducting a 6-week iron deficiency anemia study on healthy individuals,individuals with CKD, and individuals with CHF to find out if treating iron deficiency anemia with intravenous iron sucrose therapy can safely and successfully lower FGF23 levels. Iron sucrose has been shown to lower FGF23 in animal models. The short term effects of iron sucrose on FGF23 levels in CKD and CHF are not known.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Ability to understand and the willingness to sign a written informed consent.
* Iron Deficiency Anemia, as defined by
* Ferritin level < 100 ng/ml or
* Transferrin saturation <20% with ferritin 100-350 ng/ml and
* Hemoglobin < 12 g/dl

Exclusion Criteria:

* Hypersensitivity to any component of iron sucrose
* Malignancy within 5 years
* End stage renal disease or kidney transplantation
* Erythropoiesis stimulating agents
* Red blood cell transfusions within last 60 days
* Current radiotherapy or chemotherapy
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than 1.5 times normal
* Hemochromatosis
* Chronic digestive diseases
* Pregnancy or nursing
* Active alcohol or drug abuse
* Uncontrolled hypertension
* Active infection
* Hospitalization in the 4 preceding weeks
* Concomitant use of antibiotics
* Concomitant use of immunosuppression
* Inability to consent.
* Conditions, in which of the opinion of the investigator, make participation unacceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with iron deficiency anemia will be enrolled (those without CKD or HF, those with CKD only, those with HF only, and those with CKD/HF). They will be given iron sucrose as routine care for treatment of their iron deficiency anemia.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in c-terminal FGF23 measurements | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in plasma c-terminal FGF23 (RU/ml) over 6 weeks and 3 months
Change in Intact FGF23 measurements | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in plasma intact FGF23 (pg/ml) over 6 weeks and 3 months

SECONDARY OUTCOMES:
Change in Parathyroid Hormone | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Serum Parathyroid Hormone (pg/ml) over 6 weeks and 3 months
Change in Phosphate (mg/dl) | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Plasma Phosphate (mg/dl) over 6 weeks and 3 months
Change in Serum creatinine | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Serum creatinine (mg/dl) over 6 weeks and 3 months
Change in 1,25 dihydroxyvitamin D | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in 1,25 dihydroxyvitamin D (pg/ml) over 6 weeks and 3 months
Change in C-reactive protein | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in C-reactive protein (mg/L) over 6 weeks and 3 months
Change in Ferritin Measurement | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in serum ferritin (ng/ml) over 6 weeks and 3 months
Change in Iron Measurement | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Serum iron (ug/dl) over 6 weeks and 3 months
Change in Transferrin Saturation | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Transferrin Saturation (%) over 6 weeks and 3 months
Change in Hemoglobin Measurement | Weekly x 6 weeks, 1 longitudinal measurement at 3 months
  longitudinal change in Serum hemoglobin (g/dl) over 6 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rupal Mehta, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers